CLINICAL TRIAL: NCT05760365
Title: The Improvement of Medical Education by Using the Application of Three-dimensional Printing in Cardiac Catheterization
Brief Title: Three-dimensional Printing in Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FJUH110157
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Satisfaction, Personal
Keywords: 3D printed; medical education; cardiac catheterization; Heart disease
MeSH Terms: conditions — Personal Satisfaction; Heart Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slide-based presention group (Active Comparator): Received a regular learning
  Interventions: Other: Slide-based presention
- 3D-printed presention group (Experimental): Received a regular learning plus 3D printing model
  Interventions: Other: 3D printed educational model

INTERVENTIONS:
Other: 3D printed educational model — 3D printed cardiac catheterization model
  Arms: 3D-printed presention group
Other: Slide-based presention — Slide-based presention
  Arms: Slide-based presention group

SUMMARY:
Our purpose is to use 3D printing technology to make human anatomical cardiovascular model, which could apply in the medical education for medical students, in order to improve the effectiveness of the learning process to access.

DETAILED DESCRIPTION:
Background：

The medical teaching models are expansive and rare. We try to use the 3D printing technology to print cardiovascular model. By using the 3D cardiovascular model, we try to facilitate the leaning curve of understanding the cardiac catheterization.

Study Design：

This is a single-site prospective randomized controlled trial of medical education. We expect to enrolled 50 participants. Both group will receive same teaching program. Traditional education model will be used in control group, and 3D printed model will be used in the experimental group.

Methods：

We use 3D printing technology to create cardiovascular model from the CT scanning, which are drawn by professional 3D drawing staff. The students will be divided into 2 groups: the first group receive lecture/image teaching first then trained by the 3D cardiovascular model; the second group are receiving the reverse order. The satisfaction and the learning outcomes would be evaluated by the questionnaire.

Effect：

We expect the 3D cardiovascular model will bring better learning efficiency and satisfaction. Furthermore, we will construct the individual learning project by using the 3D printing model.

Key words：

3D printing, anatomy instruction, cardiovascular system, cardiac catheterization, high-fidelity simulation.

ELIGIBILITY:
Inclusion Criteria:

* Medical student, nurse practitioner and Resident in Fu Jen Catholic University Hospital

Exclusion Criteria:

* Refused to participate in the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Examination score of pre-intervention | pre-intervention
  score of pre-intervention (maximun 100 and minimum 0), higher means a better outcome
Examination score of post-intervention | immediately after the intervention
  score of post-intervention (maximun 100 and minimum 0), higher means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No